CLINICAL TRIAL: NCT01553071
Title: Phase I Trial of Intravenous Fenretinide (4-HPR) Plus Intravenous Safingol for Patients With Relapsed Malignancies
Brief Title: Phase I Trial of IV Fenretinide (4-HPR) Plus IV Safingol for Patients With Relapsed Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: drug supply issues during COVID-19
Sponsor: South Plains Oncology Consortium (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPOC-2010-002
Record Dates: First submitted 2012-03-07; First posted 2012-03-13 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Solid Tumor
Keywords: Malignancy, Relapsed; Chemotherapy, Intravenous
MeSH Terms: conditions — Neoplasms; Recurrence | interventions — Fenretinide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Investigational (Experimental): Fenretinide (4-HPR) plus Intravenous Safingol
  Interventions: Drug: Fenretinide (4-HPR) plus Intravenous Safingol

INTERVENTIONS:
Drug: Fenretinide (4-HPR) plus Intravenous Safingol — A course for this study is defined as the 5 days of treatment with Fenretinide (4-HPR) plus Safingol followed by 16 days of rest. A course is repeated every 21 days if there is no clinical evidence of disease progression for a maximum of six 5-day infusions.
  Days 1-5 of every cycle: Day 1 Fenretinide (4-HPR) intravenous emulsion: 600 mg/m2 for 24 hours Given concurrently (at the same time) with: Safingol intravenous 210 mg/m2 for 24 hours Day 2 Fenretinide (4-HPR) intravenous emulsion: 1000 mg/m2 for 24 hours Given concurrently (at the same time) with: Safingol intravenous 210 mg/m2 for 24 hours Days 3-5 Fenretinide (4-HPR) intravenous emulsion: 1000 mg/m2 continuously for 3 days Days 8 and 15 : Weekly blood draw to monitor side effects requires a clinic visit for approximately 1 hour Days 6,7,9-14, 16-21 Rest and monitor side effects.

SUMMARY:
In preclinical studies, the anti-cancer efficacy of fenretinide, a synthetic retinoid that causes cytotoxicity by mechanisms which include increased intracellular dihydroceramides, has been shown to be enhanced by safingol, a stereochemical-variant dihydroceramide precursor. This phase I study represents the first clinical trial employing this promising combination. The drug administration schedule (fenretinide given on Days 1-5, safingol given on Days 1-2 of each 21-day cycle) reflects the in vitro observation that tumor cell exposure to safingol increased fenretinide efficacy both during and after safingol administration. The total dose of fenretinide, 4600 mg/m2 over 5 days, represents a 30% total dose reduction from the single agent MTD dose of 1280 mg/m2/day x 5 days determined on the PhI-42 study. This fenretinide dose is expected to produce plasma levels in the 30?s ?M. This dose reduction has been employed to reduce the potential for overlapping hepatic toxicities between these two agents.

The administration of a reduced fenretinide dose on Day 1 (600 mg/m2 on Day 1, escalated to 1000 mg/m2/day on Days 2-5) has been selected due to earlier observations that initial exposure to the soy bean oil vehicle in the fenretinide emulsion may induce endogenous lipases, thereby permitting tolerance of higher total doses fenretinide emulsion subsequently administered. The starting dose of safingol in this study, 210 mg/m2/day x 2 days (420 mg/m2 total), corresponds to 50% of the recommended Phase II safingol dose (bolus) determined in the Schwartz, et al, Phase I study of safingol plus cisplatin 60 mg/m2 (the MTD of single-agent, intravenous (emulsion) safingol was not reached in the Phase I safingol run-in monotherapy portion of this study), and was selected to provide an adequate safety margin against the potential for overlapping toxicities (such as hepatic transaminitis).

The study has been designed to optimize the safety of this novel combination. Treatment will be administered in the inpatient setting. Central venous access will be mandated to avoid the potential for hemolysis and thrombophlebitis associated with the preclinical peripheral administration of a previous safingol formulation in rats. To reduce the incidence of hypertriglyceridemia, a revised fenretinide delivery schedule will be employed. Patients will also be encouraged to maintain a low-fat diet during fenretinide administration. Serum triglycerides will be monitored every 12 hours. To monitor for cardiac toxicity, which was noted in canine studies at the highest dose of safingol plus fenretinide tested, serum troponin T levels will be monitored daily. To limit the potential for hepatotoxicity resulting from a possible drug interaction observed between intravenous fenretinide, ceftriaxone and acetaminophen in a pediatric patient, the concurrent administration of ceftriaxone, or acetaminophen, with the fenretinide emulsion infusion will be prohibited.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria - Solid Tumor

1. Patients must have histologically or cytologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective.
2. All patients must have measurable disease documented by CT, MRI, or non-measurable disease documented by Physical Exam within 28 days prior to registration.
3. Age >18 years.
4. ECOG performance status of 0 - 2 (Karnofsky > 60%).
5. Life expectancy of greater than 3 months.
6. Patients must have adequate organ and marrow function as defined below:

   * absolute neutrophil count ≥ 1,500/μL
   * platelets ≥ 100,000/μL
   * total bilirubin ≤ 1.5 x institutional upper limit of normal (IULN)
   * AST (SGOT) ≤ 2.5 x institutional upper limit of normal (IULN) ≤ 5 x IULN for patients with liver metastases
   * ALT (SGPT) ≤ 2.5 x institutional upper limit of normal (ULN) ≤ 5 x IULN for patients with liver metastases - creatinine within institutional normal limits (WNL) OR creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
7. Effects of fenretinide and safingol on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. For women of child-bearing potential, a negative serum pregnancy test is required within 72 hours prior to receiving study drug each cycle. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
8. Ability to understand and the willingness to sign a written informed consent document.
9. Patients who have received prior treatment with oral or intravenous fenretinide as a single agent are eligible, provided they did not experience severe toxicity related to fenretinide.

Inclusion Criteria - Non-Hodgkin's Lymphoma

1. Patients must have histologically or cytologically confirmed non-Hodgkin's lymphoma for which standard therapies do not exist or are no longer effective. To be eligible for this study, lymphoma patients must have no marrow involvement as documented by routine marrow aspiration and biopsy performed within 30 days of study entry.
2. All patients must have measurable disease documented by CT, MRI, or non-measurable disease documented by Physical Exam within 28 days prior to registration.
3. Age 18 years or greater.
4. Patients must have adequate organ and marrow function as defined below:

   * Absolute neutrophil count (ANC) ≥ 1500, platelets ≥ 100,000, unless due to direct bone marrow involvement of disease.
   * Hemoglobin ≥ 8.0 gm/dL; transfusion permitted to achieve this level
   * Serum creatinine ≤ 1.5 x the upper limits of institutional normal (IULN)
   * Total bilirubin ≤ 1.5 x the IULN
   * AST/ALT ≤ 2.5 x the IULN
   * Or ≤ 5 x IULN for patients with liver metastases
5. ECOG performance status of 0 - 2 and estimated survival of at least 3 months.
6. Patients must be able to understand and agree to sign an IRB-approved informed consent form.
7. The effects of fenretinide and safingol on the developing human fetus are unknown. For this reason,women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry, for the duration of study, and for two months after study participation. For women of child-bearing potential, a negative serum pregnancy test is required within 72hours prior to receiving study drug each cycle. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
8. Patients who have received prior treatment with oral or intravenous fenretinide as a single agent are eligible, provided they did not experience severe toxicity related to fenretinide.

Exclusion Criteria:

1. Radiation therapy, chemotherapy, and other investigational agents within 3weeks (6 weeks for nitrosourea or mitomycin C) prior to starting fenretinide + safingol. Patients must have recovered from toxicities of prior therapy.
2. Concurrent administration of any other investigational agents
3. Uncontrolled intercurrent illnesses including, but not limited to, ongoing or active systemic infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, coagulation disorders; other major medical illnesses of the cardiovascular or respiratory systems or psychiatric illness/social situations that would limit compliance with study requirements.
4. Pregnant women are excluded from this study because the effects of fenretinide and safingol on the developing human fetus are unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with fenretinide and safingol, breastfeeding must be discontinued.
5. Major surgery in the last three weeks due to unknown effects of fenretinide and safingol on wound healing.
6. Patients with previously untreated brain metastases (including parenchymal, meningeal or dural-based CNS lesions) are excluded. However, patients with previously treated (surgery, radiation or both), clinically inactive brain metastases, who have not received corticosteroid therapy within three weeks of starting protocol therapy, are eligible.
7. Known allergy to egg products or soy bean oil.
8. Patients known to be HIV-positive receiving anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions.
9. Baseline fasting triglycerides > 2.5 institutional upper limit of normal (IULN) or hypertriglyceridemia requiring medication. Patients requiring medication for other dyslipidemias (i.e., elevated LDL cholesterol) are eligible.
10. Concomitant use of the following drugs (see Concomitant Medications, Section 3.3): antioxidants; herbal or other alternative therapy medications; vitamin supplements (especially vitamins A, C, and E) other than a standard dose multivitamin, acetaminophen, cyclosporine A or analogue; verapamil; tamoxifen or analogue, ketoconazole, chlorpromazine; RU486; indomethacin; or sulfinpyrazone, tetracycline, nalidixic acid, nitrofurantoin, phenytoin, sulfonamides, lithium, ceftriaxone, and amiodarone.

    If the patients discontinue usage of the above drugs, they can be eligible for enrollment into the study after a washout period of four half-lives.
11. Poorly-controlled diabetes mellitus, as defined as fasting serum glucose concentration over 200 mg/dl or a hemoglobin A1C over 7.5%.
12. Patients with an identified familial hyperlipidemia disorder.
13. Known history of allergic reactions attributed to compounds of similar chemical or biologic composition to fenretinide, such as 13-cis-retinoic acid, retinol, or all-trans-retinoic acid.
14. Patients with esophageal cancer with unresected or recurrent primary tumors in the esophagus are only permitted after discussion of patient with Study Chair due to concern of tumor necrosis and esophageal perforation.
15. Baseline (pre-treatment) serum troponin T (TnT) ≥ 0.03 ng/mL. Troponin T levels may be rechecked and therapy given if levels decrease to < 0.03 ng/mL.
16. Baseline (pre-treatment) EKG with any of the following changes consistent with cardiac ischemia:

    * significant ST depression (ST depression of ≥2 mm, measured from isoelectric line to the ST segment at a point 60 msec from the end of the QRS complex)
    * significant ST elevation (> 1mm in limb lead or 2 mm in precordial lead measured at a point 0.04 sec (1 mm) after the J-point [the end of the QRS complex] and compared to baseline [line drawn from P start to T end])

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-11; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose of an intravenous safingol in combination with fenretinide | approximately six months
  The primary outcome mesure of this study is to determine the maximum tolerated dose (MTD) of an intravenous (emulsion) safingol when administered as a continuous intravenous (c.i.v.) infusion for two days, once every 3 weeks, in combination with fenretinide (4-HPR) intravenous emulsion administered as a continuous intravenous infusion for five days, once every 3 weeks.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Texas Southwestern, Dallas, Texas
  - Joe Arrington Cancer Center/Covenant Children's Hospital, Lubbock, Texas
  - University Medical Center, Lubbock, Texas

REFERENCES:
- [Derived] Boulter AC, Maurer BJ, Pogue M, Kang MH, Cho H, Knight A, Reynolds CP, Quick D, Awasthi S, Gerber DE. Phase I trial of intravenous fenretinide (4-HPR) plus safingol in advanced malignancies. Cancer Chemother Pharmacol. 2023 Aug;92(2):97-105. doi: 10.1007/s00280-023-04543-6. Epub 2023 May 18. PMID 37199745
- [Derived] Cho HE, Maurer BJ, Reynolds CP, Kang MH. Hydrophilic interaction liquid chromatography-tandem mass spectrometric approach for simultaneous determination of safingol and D-erythro-sphinganine in human plasma. J Chromatogr B Analyt Technol Biomed Life Sci. 2019 Apr 1;1112:16-23. doi: 10.1016/j.jchromb.2019.02.023. Epub 2019 Feb 22. PMID 30836314